CLINICAL TRIAL: NCT04490642
Title: Linguistic Validation of the Childhood Bladder and Bowel Dysfunction Questionnaire (CBBDQ) for 5-12 Years Old in Korean
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Kwanjin Park, Associate Professor, Seoul National University Hospital
Other Study IDs: 2006-203-1137
Record Dates: First submitted 2020-07-26; First posted 2020-07-29 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Dysfunctional Voiding; Bladder Dysfunction; Bowel Dysfunction; Pediatric Urology
MeSH Terms: conditions — Intestinal Diseases | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Concomitant bladder and bowel Dysfunction: 25 patients with concomitant bladder and bowel dysfunction.
  Interventions: Other: Questionnaire
- Those without concomitant bladder and bowel dysfunction: 25 patients without concomitant bladder and bowel dysfunction.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Final version Childhood Bladder and Bowel Dysfunction for 5-12 years old questionnaire in Korean language to patients who never encountered beforehand in other available languages (Dutch, English).

SUMMARY:
The study is to conduct a linguistic and cultural validation of the Children Bladder and Bowel Dysfunction (CBBDQs) for 5-12 years old from English to Korean. Once it has been validated into the Korean language, it will be a valuable source that will better serve patients with BBD symptoms in an outpatient setting and use in future clinical studies.

DETAILED DESCRIPTION:
BBD, or Bladder and Bowel Dysfunction, is relatively a common disorder affecting approximately 40% of children, it has significant and detrimental effects on patients such as decreased quality of life, psychosocial distress, and recurrent vesicoureteral reflux (VUR) accompanied by Urinary Tract Infection (UTI). A study has found that a large number of BBD patients have comorbid neuropsychiatric disorders such as Attention Deficit Hyperactive Disorders (ADHD) and Obsessive-Compulsive Disorder (OCD). Furthermore, neuropsychiatric patients with concomitant dysfunctional voiding have significantly less favorable outcomes both physically and psychologically than those with BBD only.

With a wide range of life-debilitating symptoms and outcomes, a combination of bladder and bowel dysfunction is often missed or unrecognized by caregivers and clinicians. Some patients do not outgrow as they age, and symptoms continue into adulthood. Moreover, recurrent VUR and UTI due to dysfunctional voiding may lead to kidney failure and renal scarring.

In order to assist with diagnosing bladder and bowel dysfunction, valid questionnaires are needed. However, to this present day, there is no gold standard questionnaire that assesses concomitant dysfunctions. Some questionnaires ask the guardians to fill out on behalf of the patients, which can be perplexing in evaluating symptoms as patient- and parents- reported symptoms are different.

The Children Bladder and Bowel Dysfunction Questionnaire (CBBDQs) for 5-12 years old was originally developed by van Engeleburg-van Lonkhuyzen M. et al., and is age-specific and appropriate 18 items that both measures bladder and bowel dysfunction. It adhered COSMIN (COnsensus- Based Standards for the selection of health Measurement Instruments), and has been proven to be easy to fill out and suitable to be completed by either patients or caregivers. Most importantly, it allows professionals to evaluate the symptoms effectively. To best of our knowledge, it has not been translated into other languages than English (from the original language, Dutch). As it is only available in English and Dutch, linguistic and cultural validations are necessary as there is no similar questionnaire in Korean.

This study followed systematic guidelines outlined by COSMIN (COnsensus-based Standards for the selection of health Measurement Instruments) and similar to the linguistic validation (development) of the Korean version of the Dysfunctional Voiding Symptoms Score (DVSS) by Park et al.

The study aims to conduct a linguistic and cultural validation of the Children Bladder and Bowel Dysfunction (CBBDQs) for 5-12 years old from English to Korean. Once it has been validated into the Korean language, it will be a valuable source that will better serve patients with BBD symptoms in an outpatient setting and use in future clinical studies.

ELIGIBILITY:
Inclusion Criteria:

* Those with or without bladder and bowel dysfunction.
* Between the ages of 5 to 12 years old.

Exclusion Criteria:

- Younger than 5 years and older than 12 years of age.

Ages: 5 Years to 12 Years | Sex: All
Age Groups: Child
Study Population: A total of 50 subjects (25 subjects with bladder and bowel dysfunction and 25 without) will be recruited from the outpatient unit of pediatric urology.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-07-27 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
CBBDQs Score | 1 day
  Measured score of the Childhood Bladder and Bowel Dysfunction Questionnaire for 5-12 years old.

CONTACTS AND LOCATIONS:
Overall Officials: Kwanjin Park, M.D. Ph.D, Study Chair — Seoul National University Hospital
Locations (2):
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - Seoul National University Children's Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No